CLINICAL TRIAL: NCT02549859
Title: Long-term Effect of Low Frequency 60Hz Stimulation on Aspiration, Freezing of Gait and Other Axial and Motor Symptoms in PD Patients With Bilateral STN DBS
Brief Title: Long-term Effect of Low Frequency Stimulation on Aspiration and Freezing of Gait in PD With STN DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 15-0539
Record Dates: First submitted 2015-08-31; First posted 2015-09-15 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease
Keywords: DBS; Low frequency stimulation; Dysphagia; Freezing of gait
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (DBS) (Experimental): All patients were treated and assessed under three conditions (60 Hz DBS, 130 Hz DBS and no DBS) at Visit 1 (V1), were then treated with 60 Hz DBS for at least 6 months (14.5 months on average), and were finally reassessed during a second visit (V2) under the same three conditions as V1. The order of treatment/assessment under the three conditions was randomized at each visit.
  Interventions: Device: Deep Brain Stimulation (DBS) at 60 Hz; Device: Deep Brain Stimulation (DBS) at 130 Hz; Device: Deep Brain Stimulation (DBS) Off (Sham)

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) at 60 Hz — Bilateral subthalamic nucleus deep brain stimulation at 60 Hz
  Other Names: Low Frequency Stimulation (LFS)
Device: Deep Brain Stimulation (DBS) at 130 Hz — Bilateral subthalamic nucleus deep brain stimulation at 130 Hz
  Other Names: High Frequency Stimulation (HFS)
Device: Deep Brain Stimulation (DBS) Off (Sham) — Deep Brain Stimulation (DBS) Off (Sham)

SUMMARY:
Our recent study (Xie et al, Neurology 2015; 84: 415-420) found that bilateral STN DBS of 60Hz, compared to the traditional 130Hz, decreased the aspiration frequency and swallowing difficulty, freezing of gait (FOG), and other axial symptoms and parkinsonism in Parkinson patients with FOG refractory to 130Hz and medications. The benefit of 60Hz stimulation persisted during the 6-week study period, but with worsening tremor in one patient. However, it remains unknown whether the benefit of 60Hz would persist on prolonged stimulation period, and whether there is carry-over effect across different conditions. Hence, the investigators would like to test the hypothesis that the 60Hz stimulation, compared to 130Hz might have persistent benefit over an extended period in reducing the swallowing dysfunction, FOG, and other axial symptoms in these PD patients even after correcting the potential carry-over effect.

DETAILED DESCRIPTION:
The investigators will enroll 14 Parkinson patients with bilateral STN DBS and refractory FOG to 130Hz stimulation and dopaminergic medications for two visits of at least 6-month apart. The 6 patients remaining on 60Hz stimulation after our previous study consisting of 7 patients will be assessed once again as visit-2 after previous visit-1 of their last study. We anticipate to have 20 patents complete for visit-1 and at least 18 patients complete for visit-2 in this randomized double-blind prospective crossover study with their usual medication "on" state, with 6-7 patients on each starting condition (60Hz vs 130Hz vs DBS off). Swallowing function on modified barium swallowing test and swallowing questionnaire, FOG in stand-walk-sit test and questionnaire, and other axial and motor function on UPDRS-III will be assessed under each DBS condition. Changes in measurements between 60Hz and 130Hz at each visit and under 60Hz between two visits will be analyzed, with swallowing function and FOG as primary, and the rest as secondary outcomes, correcting for potential carryover effect. Changes between other DBS conditions might also be explored in this 2-year study.

This would be the first study on the long-term effect of 60Hz stimulation on dysphagia, FOG and other axial and motor symptoms in Parkinson patients with bilateral STN DBS and FOG refractory to 130Hz stimulation and dopaminergic medications, which will have significant impact on the treatment of difficult axial symptoms of high morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* PD patients with bilateral STN DBS placement and FOG at 130Hz even at usual medication "on" state.

Exclusion Criteria:

* Known history of recent aspiration pneumonia

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xie, MD PhD, Principal Investigator — Department of Neurology, University of Chicago
Locations (1):
- University of Chicago, Department of Neurology, Chicago, Illinois, United States

REFERENCES:
- [Result] Xie T, Vigil J, MacCracken E, Gasparaitis A, Young J, Kang W, Bernard J, Warnke P, Kang UJ. Low-frequency stimulation of STN-DBS reduces aspiration and freezing of gait in patients with PD. Neurology. 2015 Jan 27;84(4):415-20. doi: 10.1212/WNL.0000000000001184. Epub 2014 Dec 24. PMID 25540305
- [Result] Xie T, Bloom L, Padmanaban M, Bertacchi B, Kang W, MacCracken E, Dachman A, Vigil J, Satzer D, Zadikoff C, Markopoulou K, Warnke P, Kang UJ. Long-term effect of low frequency stimulation of STN on dysphagia, freezing of gait and other motor symptoms in PD. J Neurol Neurosurg Psychiatry. 2018 Sep;89(9):989-994. doi: 10.1136/jnnp-2018-318060. Epub 2018 Apr 13. PMID 29654112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 patients were screened for eligibility at a hospital-associated specialty clinic in Chicago, IL.
Pre-assignment Details: Eleven of 15 screened participants were enrolled; four did not meet inclusion/exclusion criteria. Five of the enrolled participants had participated in a previous study and had been treated on 60Hz DBS since then; their Visit 1 (V1) measurements were taken from the previous study.
Period: Visit 1
Arm/Group | Deep Brain Stimulation (DBS)
Started | 11
Completed | 11
Not Completed | 0
Period: Long-term 60 Hz DBS
Arm/Group | Deep Brain Stimulation (DBS)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Study Closed | 1
Period: Visit 2
Arm/Group | Deep Brain Stimulation (DBS)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deep Brain Stimulation (DBS)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 6
  Asian | 1
  Black | 0
  Hispanic or Latino | 4
Region of Enrollment [Number; unit: participants]
  United States | 11
Parkinson's Disease Duration [Mean (Standard Deviation); unit: years] | 14.2 (5.7)
DBS at High Frequency Stimulation Duration [Mean (Standard Deviation); unit: years] | 3.5 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Aspiration Events on Videofluoroscopic Swallow Study at Visit 1
Description: A speech pathologist used the Penetration-Aspiration Scale (PAS) to rate swallows captured by a radiologist during VFSS recording. PAS is an 8-point interval scale: a score of 0 indicates no penetration or aspiration & a score of 6-8 indicates aspiration of increasing severity. For the purpose of this study, aspiration was dichotomized to "0" if PAS score was under 6 or "1" if PAS score was between 6-8. Frequency of aspiration events was calculated by adding number of aspiration events in VFSS under various liquid & food textures. The maximum aspiration frequency was 12 if aspiration occurred on every texture after 2 trials. Lower aspiration frequency means better swallowing function.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- DBS 60Hz: Participants were on DBS 60Hz for at least 30 min before evaluation. The order of administration of DBS conditions was randomized, and the participants and study team were blinded to the DBS condition.
- DBS 130Hz: Participants were on DBS 130Hz for at least 30 min before evaluation. The order of administration of DBS conditions was randomized, and the participants and study team were blinded to the DBS condition.
- DBS Off: Participants were on DBS off for at least 30 min before evaluation. The order of administration of DBS conditions was randomized, and the participants and study team were blinded to the DBS condition.
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 0.6 (0.8) | 2.9 (2.1) | 1.2 (1.7)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

2. Primary Outcome: Perceived Swallowing Difficulty on Swallowing Disturbance Questionnaire at Visit 1
Description: The Swallowing Disturbance Questionnaire contains 15 items. Each item has 4-points ranging from 0 (absence of symptoms) to 3 (severe or very frequent). Total score ranges from 0-45, with higher scores corresponding to more severe swallowing disturbance.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 1.1 (1.0) | 3.3 (2.1) | 3.1 (1.9)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.01, Paired t-test, 2 sided

3. Primary Outcome: Freezing of Gait Questionnaire at Visit 1
Description: The Freezing of Gait (FOG) Questionnaire contains 6 items to evaluate the severity of FOG in patients with Parkinson's disease. Each item has 5 points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-24, with higher scores corresponding to more severe FOG.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 3.0 (3.7) | 9.3 (4.1) | 5.1 (3.8)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.01, Paired t-test, 2 sided

4. Primary Outcome: Stand-Walk-Sit Freezing of Gait Spells at Visit 1
Description: The Stand-Walk-Sit (SWS) Test assesses freezing of gait (FOG) spells observed when standing up, walking 7 meters, and returning to a seated position. The greater the number of FOG spells counted, the worse the FOG symptoms.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 0.1 (0.2) | 3.0 (3.8) | 1.6 (1.6)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

5. Primary Outcome: Stand-Walk-Sit Time at Visit 1
Description: Stand-Walk-Sit (SWS) Time measures the total time taken to complete the SWS test of standing up, walking 7 meters, and returning to a sitting position. The longer time (in seconds) it took to complete the SWS test, the worse the FOG symptoms.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
seconds | 22.1 (7.1) | 28.5 (8.5) | 23.6 (6.0)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

6. Primary Outcome: Frequency of Aspiration Events on Videofluoroscopic Swallow Study at Visit 2
Description: as for outcome 1
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 2.0 (2.4) | 3.0 (2.5) | 2.4 (2.6)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

7. Primary Outcome: Perceived Swallowing Difficulty on Swallowing Disturbance Questionnaire at Visit 2
Description: as for outcome 2
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 4.8 (6.9) | 7.4 (8.9) | 5.7 (6.9)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

8. Primary Outcome: Freezing of Gait Questionnaire at Visit 2
Description: as for outcome 3
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 5.9 (4.4) | 11.2 (4.1) | 7.0 (4.0)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.01, Paired t-test, 2 sided

9. Primary Outcome: Stand-Walk-Sit Freezing of Gait Spells at Visit 2
Description: as for outcome 4
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 2.2 (3.8) | 6.1 (7.0) | 2.5 (2.8)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

10. Primary Outcome: Stand-Walk-Sit Time at Visit 2
Description: as for outcome 5
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
seconds | 26.5 (12.2) | 38.4 (26.0) | 27.8 (11.9)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

11. Secondary Outcome: Unified Parkinson's Disease Rating Scale-III Total Score at Visit 1
Description: Unified Parkinson's Disease Rating Scale-III (UPDRS-III) contains 33 items. Each item has 5-points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-132, with higher scores corresponding to more severe parkinsonism.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 22.8 (10.4) | 33.7 (8.3) | 34.4 (12.1)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.01, Paired t-test, 2 sided

12. Secondary Outcome: Axial Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 1
Description: The axial subscore of Unified Parkinson's Disease Rating Scale-III (UPDRS-III) contains 7 items. Each item has 5-points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-28, with higher scores corresponding to more severe axial symptoms. Specifically, axial symptoms include: speech, facial expression, arising from chair, gait, freezing of gait, postural stability, posture.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 3.8 (3.3) | 8.9 (3.4) | 6.9 (4.4)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.001, Paired t-test, 2 sided

13. Secondary Outcome: Bradykinesia Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 1
Description: The bradykinesia subscore of Unified Parkinson's Disease Rating Scale-III (UPDRS-III) contains 11 items. Each item has 5-points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-44, with higher scores corresponding to more severe bradykinesia. Specifically, bradykinesia symptoms include: finger tapping right hand, finger tapping left hand, hand movements right hand, hand movements left hand, pronation-supination movements right hand, pronation- supination movements left hand, toe tapping right foot, toe tapping left foot, leg agility right leg, leg agility left leg, global spontaneity of movement.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 11.7 (5.3) | 16.6 (4.6) | 17.1 (5.0)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

14. Secondary Outcome: Rigidity Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 1
Description: The rigidity subscore of Unified Parkinson's Disease Rating Scale-III (UPDRS-III) contains 5 items. Each item has 5-points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-20. with higher scores corresponding to more severe rigidity. Specifically, rigidity symptoms include: rigidity neck, rigidity right upper extremity, rigidity left upper extremity, rigidity right lower extremity, rigidity left lower extremity.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 4.0 (2.4) | 4.9 (2.5) | 6.0 (3.1)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

15. Secondary Outcome: Tremor Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 1
Description: The tremor subscore of Unified Parkinson's Disease Rating Scale (UPDRS-III) contains 10 items. Each item has 5-points ranging from 0 (absence of symptoms) to 4 (severe). Total score ranges from 0-40, with higher scores corresponding to more severe tremor. Specifically, tremor symptoms include: postural tremor right hand, postural tremor left hand, kinetic tremor right hand, kinetic tremor left hand, rest tremor amplitude right upper extremity, rest tremor amplitude left upper extremity, rest tremor amplitude right lower extremity, rest tremor amplitude left lower extremity, rest tremor amplitude lip/jaw, constancy of rest tremor.
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 11 | 11 | 11
score on a scale | 1.8 (2.2) | 1.2 (2.1) | 2.5 (3.4)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

16. Secondary Outcome: Unified Parkinson's Disease Rating Scale-III Total Score at Visit 2
Description: as for outcome 11
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 27.1 (9.1) | 32.4 (7.1) | 31.4 (10.1)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

17. Secondary Outcome: Axial Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 2
Description: as for outcome 12
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 6.8 (4.7) | 10.4 (3.9) | 8.1 (4.0)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

18. Secondary Outcome: Bradykinesia Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 2
Description: as for outcome 13
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 12.8 (3.5) | 16.3 (2.3) | 15.7 (3.7)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p < 0.05, Paired t-test, 2 sided

19. Secondary Outcome: Rigidity Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 2
Description: as for outcome 14
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 4.3 (2.2) | 3.8 (2.1) | 4.8 (2.4)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

20. Secondary Outcome: Tremor Subscore of Unified Parkinson's Disease Rating Scale-III at Visit 2
Description: as for outcome 15
Time Frame: Immediately following treatment for at least 30 minutes
Population: Participants completing Visit 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
Number analyzed (Participants) | 10 | 10 | 10
score on a scale | 1.6 (2.6) | 0.2 (0.7) | 1.2 (2.0)
Statistical Analysis 1: Comparison: DBS 60Hz vs DBS 130Hz; Test type: Superiority; p > 0.05, Paired t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected beginning from the time of consent and extending until all study procedures were complete for the patient, an average of 14.5 months. After patient's second visit was completed, no further AEs were collected.
Description: AE and SAE were defined by the investigator as any medical event that the patient and doctor considered medically relevant.
Arm/Group | DBS 60Hz | DBS 130Hz | DBS Off
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
It is only tested on PD patients with FOG refractory to the 130Hz of bilateral STN DBS at usual medication "on" state, with limited participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02549859/Prot_SAP_000.pdf